CLINICAL TRIAL: NCT03173885
Title: An RCT Evaluating the Implantation Potential of Vitrified Embryos Screened by Next Generation Sequencing Following Trophectoderm Biopsy, Versus Vitrified Unscreened Embryos in Good Prognosis Patients Undergoing IVF
Brief Title: Investigating the Cryopreserved Blastocyst's ImplantatiOn Potential After Genetic Screening
Acronym: BIOPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the slow recruitment of patients
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B670201629937; 2016/1235 (Other: Ghent University Hospital)
Record Dates: First submitted 2017-05-19; First posted 2017-06-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Infertility; Preimplantation Genetic Screening
MeSH Terms: conditions — Infertility | interventions — Preimplantation Diagnosis

STUDY DESIGN:
Intervention Model Description: RCT (randomized controlled trial)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PGS (genetic screening) (Experimental): Intent to transfer single cryopreserved embryo, selection based on euploid status (after preimplantation genetic screening) and standard morphological assessment
  Interventions: Diagnostic Test: Preimplantation Genetic Screening
- no PGS (no genetic screening) (No Intervention): Intent to transfer single cryopreserved embryo, selection based on standard morphological assessment

INTERVENTIONS:
Diagnostic Test: Preimplantation Genetic Screening — * laser assisted hatching
  * trophectoderm biopsy
  * next generation sequencing
  Arms: PGS (genetic screening)

SUMMARY:
This is a two-arm parallel group randomized controlled trial at the Department of Reproductive Medicine at Ghent University Hospital. Women >=18 and <37 years of age undergoing their first or second IVF/ICSI treatment, with at least 2 good quality blastocysts remaining after fresh embryo transfer will be randomized to either transfer of a cryopreserved blastocyst selected based on morphology (standard treatment arm) or transfer of a cryopreserved blastocyst selected based on PGS and morphology (intervention treatment arm).

ELIGIBILITY:
Inclusion Criteria:

* at least 2 blastocysts suitable for biopsy on day 5 of embryo development remaining after fresh transfer
* willing and able to give informed consent
* infertility as an indication for IVF/ICSI
* first or second IVF/ICSI cycle
* patients willing to accept single embryo transfer
* BMI range 18 to 35 kg/m2

Exclusion Criteria:

* any type of genetic abnormality or family history of genetic abnormality in subject or partner
* any other non-study related preimplantation genetic testing
* three or more clinical miscarriages (recurrent pregnancy loss, RPL)
* recurrent implantation failure (RIF): no positive β-hCG after transfer (fresh IVF/ICSI cycle or frozen) with no less than 6 cleavage stage embryos or no less than 4 blastocysts, all of good quality and of appropriate developmental stage
* severe endometriosis
* abnormal uterine cavity
* cycles requiring surgical sperm recovery procedures, total asthenozoospermia and/or globozoospermia
* treatment involving use of donor oocytes or use of gestational carrier

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | At 7 - 8 gestational weeks
  Rate of clinical pregnancy (a pregnancy diagnosed by ultrasonic visualisation of one or more gestational sacs with fetal heart beat) after transfer of embryo in PGS arm versus in no PGS arm.

SECONDARY OUTCOMES:
Biochemical pregnancy | At 7 -8 gestational weeks
  Rate of biochemical pregnancy (a pregnancy diagnosed only by either serum or urine β-hCG, and the serial results decrease to negative; no ultrasonic visualisation of one or more gestational sacs) after transfer of embryo in PGS arm versus in no PGS arm.
Clinical miscarriage | At 7 - 16 gestational weeks
  Rate of clinical miscarriage (intrauterine pregnancy demise confirmed by ultrasound or histology) after transfer of embryo in PGS arm versus in no PGS arm.
Live birth | At delivery
  Rate of live birth (> 24 weeks gestation) after transfer of embryo in PGS arm versus in no PGS arm.
Aneuploidy | At delivery
  Rate of aneuploid versus rate of euploid embryos in PGS arm.

CONTACTS AND LOCATIONS:
Overall Officials: Petra De Sutter, M.D; PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital - Department of Reproductive Medicine, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291